CLINICAL TRIAL: NCT04399096
Title: Sound and Vision: A Collaboration Between Service-users, Artists and the Public to Explore the Lived Experience of Hallucinations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Cambridgeshire and Peterborough NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, John Suckling, Director of Research in Psychiatric Neuroimaging, University of Cambridge
Other Study IDs: 269849
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Parkinson Disease; Hallucinations
Keywords: hallucination
MeSH Terms: conditions — Schizophrenia; Parkinson Disease; Hallucinations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population: The general public attending exhibitions of the artworks who wish to complete the on-line questionnaire and feedback

SUMMARY:
Sound and Vision: A collaboration between service-users, artists and the public to explore the lived experience of hallucinations

DETAILED DESCRIPTION:
Sound and Vision will pair local artists with patients who have had hallucinations to create art pieces that represent their hallucinatory experiences. Patients with diagnoses of schizophrenia and Parkinson's disease will be invited to take part in participating National Health Service (NHS) clinics, to capture and compare a wide range of hallucinatory experiences. Patients will meet with artists on several occasions who will then develop the piece, which may be a painting, drawing, or other media that the artist and service-user jointly select.

Completed artworks will be the centrepiece for an exhibition at United Kingdom (UK) science festivals and a digital (on-line) presentation. The exhibition will be accompanied by researchers explaining the brain science of hallucinations, recordings of patients and artists describing their experience with hallucinations and the process of developing the artworks, booklets cataloguing the exhibition, and art materials available for artistic expression of their own experiences. A digital compendium of the artworks and supporting material will be publicly available alongside the opportunity to complete an online survey exploring the themes of the artworks and collecting information on personal experiences. The objectives are to engage the public in an appreciation of the experience of hallucinations and their prevalence across many common mental health and neurodegenerative disorders, as well as an experience many people will share without ever being diagnosed. The exhibition will also encourage the public to share their own experiences through the online questionnaires creating a platform to begin to improve the understanding of the diversity of hallucination-like experiences in the general population.

ELIGIBILITY:
No particular inclusion or exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The general publication attending an exhibition of artworks depicting the experience of hallucinations.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
University of Miami Parkinson's disease Hallucinations Questionnaire (UM-PDHQ) | Through study completion, an average of 1 year
  The University of Miami Parkinson's disease Hallucinations Questionnaire (UM-PDHQ) is composed of 6 quantitative and 14 qualitative items to define the key characteristics of hallucinations in Parkinson's Disease. The first 6 questions score the severity of hallucinations with a minimum score is zero and a maximum of 14, with greater score indicating greater severity. The remaining 14 questions have qualitative answers.
The Multi-Modality Unusual Sensory Experiences Questionnaire (MUSEQ) | Through study completion, an average of 1 year
  The Multi-Modality Unusual Sensory Experiences Questionnaire (MUSEQ) is a 43-item self-report measure with each item rated on a five-point Likert scale, and assesses unusual sensory experiences in six modalities: auditory, visual, olfactory, gustatory, bodily sensations, and sensed presence. The minimum score is zero, the maximum score is 173 with a greater score indicating a higher frequency of unusual sensory experiences.

CONTACTS AND LOCATIONS:
Overall Officials: John Suckling, Principal Investigator — University of Cambridge; Emilio Fernandez-Egea, Principal Investigator — Cambridgeshire and Peterborough NHS Foundation Trust; James Rowe, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Cambridge and Peterborough NHS Trust, Cambridge, Cambs
  - Cambridge University Hospital, Cambridge, Cambs

REFERENCES:
- [Background] Rollins CPE, Garrison JR, Simons JS, Rowe JB, O'Callaghan C, Murray GK, Suckling J. Meta-analytic Evidence for the Plurality of Mechanisms in Transdiagnostic Structural MRI Studies of Hallucination Status. EClinicalMedicine. 2019 Feb 21;8:57-71. doi: 10.1016/j.eclinm.2019.01.012. eCollection 2019 Feb. PMID 31193632